CLINICAL TRIAL: NCT02665520
Title: Phase 1 Study of the Use of Autologous Penile Stem Cells in Men With Erectile Dysfunction
Brief Title: Penile Intracavernosal Stem Cells Therapy for Erectile Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elaj medical centers (Other)
Collaborators: King Saud University (Other)
Responsible Party: Principal Investigator, Mohamad Habous, Dr Mohamad Habous, Elaj medical centers
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Elaj stem cells 1
Record Dates: First submitted 2015-03-09; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Erectile Dysfunction
Keywords: stem cells injections; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cells injection in penis (Active Comparator): Treatment Injection of adipose derived cells into penis experimental;randomised
  Interventions: Procedure: liposuction for retrieval of own stem cells from fat cells
- controled arm (No Intervention)

INTERVENTIONS:
Procedure: liposuction for retrieval of own stem cells from fat cells
  Arms: stem cells injection in penis

SUMMARY:
Autologous Fat Derived Stem Cell treatment of ED.

To assess safety and primary efficacy of stem cell infusion in refractory ED.

To investigate the success rate and durability of success of using this new therapy in management of moderate and sever cases of erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Male 40 years old and older suffering from moderate to sever erectile dysfunction -

Exclusion Criteria:

* Inability to give informed consent or attend follow up
* Severe diabetic neuropathy (to be defined ? Charcot joints, diabetic ulcers?) or other neuropathic disease
* Viral disease from infectivity viewpoint
* Major penile fibrosis or severe Peyronie's disease
* Severe primary large vessel ED (defined as PSV less than 15cm/s after ICI)
* Severe primary venous leakage ED (defined as EDV more than 10cm/s after ICI)
* Prior systemic chemotherapy, or radiotherapy to donor or recipient area
* Not in potentially active sexual relationship
* Age less than 40 or over 70

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events that occur during or after the procedure to measure safety and tolerability | 1 year
  to assess efficacy and safety of injection of stem autologous stem cells in penis of ED patients

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Binsaleh, MD, Study Director — King Saud University
Locations (2):
- Saudi Arabia (2):
  - Elaj medical group, Jeddah, Outside U.S./Canada
  - kING SAUD UNIVERSITY, Riyadh